CLINICAL TRIAL: NCT03635554
Title: Translation and Clinical Implementation of a Test for Language and Short-term Memory in Aphasia
Brief Title: Translation and Clinical Implementation of a Test of Language and Short-term Memory in Aphasia
Acronym: ClinTALSA
Status: Enrolling by invitation | Type: Observational
Sponsor: Temple University (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Nadine Martin, Professor Communication Sciences and Disorders, Temple University
Other Study IDs: TempleU2
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Aphasia
Keywords: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to develop a clinically feasible version of a laboratory-developed assessment battery for language and verbal short-term memory difficulties in aphasia.

DETAILED DESCRIPTION:
Over five years, we will develop a clinically feasible test that can be used to assess in-depth the language and verbal short-term memory abilities of individuals with aphasia (Called the TALSA - Temple Assessment of Language and Short-term memory in Aphasia. Based on a test that we have developed and tested over the past decade, we will create a shorter version that can be used by clinicians in a rehabilitation setting. The data to support this development will come from two sources: (1) clinicians in rehabilitation facilities who will use the new clinical test and provide feedback on the test (administration, value etc) and (2) people with aphasia who will be administered the longer version to help us identify the best test items in the laboratory version of the TALSA to be carried over to the shorter clinical version.

We are recruiting individuals with aphasia as well as people without aphasia (to serve as controls) to help with development of this assessment battery. The battery consists of between 15 and 20 subtests that assess many aspects of language and verbal short-term memory.

ELIGIBILITY:
Inclusion Criteria:

* . single or multiple left hemisphere lesions
* at least one year post-stroke.
* high-school educated
* negative histories for mental illness and alcohol/substance abuse.
* passed an audiometric pure-tone, air conduction screening at 25 dB HL at 1K, 2K and 4K Hz for at least one ear.

Exclusion Criteria:

English as a second language Right hemisphere stroke Less than 6 months post-onset of stroke.

Ages: 21 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with aphasia will have single or multiple left hemisphere lesions, but no right hemisphere lesions. They can be between the ages of 21 and 80. Their aphasia can range in severity from mild to severe and can be of any type except global aphasia. Their language output can be fluent or nonfluent and their comprehension can be mild moderately impaired.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportions correct on subtests of the Test of Language and Short-term Memory in Aphasia (TALSA) | two to three years December 1, 2017 through December 15, 2017 through November 30, 2022.
  Participants will be administered 15-20 subtests of the TALSA that assess aspects of language (phoneme discrimination, sentence comprehension) and short-term memory (e.g., repetition span) abilities. Their responses on these measures will be evaluated in a item response analysis to determine which items are ideal to use in a smaller version of this test that is feasible to use in clinical practice. Another group of people with aphasia will be administered the clinical version (when it is complete) to develop normative data for that assessment battery.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Martin, Ph.D., Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States